CLINICAL TRIAL: NCT03207568
Title: RE-GENERATION: An EU Clinical Study to Evaluate the Safety and Performance of the Relay Pro and Relay Non Bare Stent (NBS) Pro Stent-graft Devices in Patients With Thoracic Aortic Pathologies
Brief Title: RE-GENERATION: The Safety and Performance of the Relay Pro and Relay NBS Pro Stent-graft Devices in the European Union (EU)
Acronym: RE-GENERATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bolton Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-0011-14
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Aorta, Thoracic Pathologies; Aortic Aneurysm, Thoracic; Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aortic Aneurysm | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Intervention Model Description: Relay Pro and Relay NBS Pro device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relay Pro Device (Experimental): The Relay Pro thoracic stent-graft will be used to treat pathologies eligible for thoracic endovascular aortic repair (TEVAR).
  Interventions: Device: Thoracic Endovascular Aortic Repair (TEVAR)

INTERVENTIONS:
Device: Thoracic Endovascular Aortic Repair (TEVAR) — thoracic endovascular repair (TEVAR) with a thoracic stent-graft
  Other Names: RELAY PRO STENT GRAFT; RELAY NBS PRO STENT GRAFT

SUMMARY:
The objective of the study is to evaluate the safety and performance of Relay Pro and Relay NBS Pro devices in humans having thoracic aortic pathologies.

Clinical results will be used to apply for the CE certification.

DETAILED DESCRIPTION:
This is a prospective, multicenter, non-randomized, single arm clinical study in patients presenting thoracic aortic pathologies. Patients with thoracic aortic pathologies who are planned to undergo thoracic endovascular aortic repair (TEVAR) with a stent-graft based on routine clinical assessments performed as part of the patients' standard care will be screened after obtaining the informed consent from the patients, and if eligible, enrolled and scheduled for the implantation procedure with the study device.

Following a baseline assessment, the implantation procedure will be performed according to the Instructions for Use and local routine practice. A follow-up visit will be performed 30 days after the implantation procedure. The investigator will perform assessments of the implantation procedure and device system and document adverse events and device deficiencies.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with thoracic aorta pathology (aneurysm, pseudoaneurysm, dissection, penetrating ulcer or intramural hematoma) suitable for TEVAR with a Relay Pro or Relay NBS Pro stent-graft; diagnosis must be confirmed by contrast computed tomography angiography (CTA) or magnetic resonance imaging (MRI) within 3 months of the planned implant procedure.
* Proximal and distal aortic necks suitable for stent-graft placement (i.e., diameter ranging between 18 and 42 mm)
* Proximal and distal landing zones suitable for the stent-graft
* Adequate vascular access for insertion of the delivery system, i.e., femoral or iliac arteries a minimum 6 mm in diameter to accommodate the 19 to 22-Fr outer-diameter delivery system and no excessive disease precluding delivery system entry/passage or iliac arteries that could be extended via an access conduit.
* Written informed consent provided by the subject him/herself (not a representative) upon enrollment

Exclusion Criteria:

Patients who meet one or more of the following criteria are not eligible:

* Aneurysm/lesion location not accessible to the delivery system and stent placement
* Arterial access size insufficient for delivery system entrance or impossibility to perform a surgical access conduit
* Treatment of lesion that would require a delivery system with usable length greater than 90 cm
* Excessive arterial disease precluding delivery system entrance or passage
* Systemic infection
* Arterial tortuosity not allowing passage of the delivery system
* Arterial or aneurysm/lesion size incompatible with stent graft
* Has congenital connective tissue disease rendering the aneurysm/lesion untreatable
* Mycotic aneurysm/lesions
* Aortic inner diameter that cannot accommodate the expanded Inner Secondary Sheath outer diameter of approximately 10mm
* Native bleeding diathesis
* Any condition (medical or anatomic) which makes the patient not suitable for endovascular
* repair according to the opinion of the investigator
* Untreatable allergy or history of allergic reaction to radiographic contrast medium
* Untreatable allergy or history of allergic reaction to anticoagulants
* Hypersensitivity to polyester or nitinol or any of the components of the Relay device
* Patient underwent prior thoracic aortic repair (endovascular or surgical)
* Participation in an investigational clinical study involving a new chemical entity or medical device within 3 months or 1 year, respectively, prior to the planned procedure
* Patient not willing to give consent for transmission of personal "pseudonymised" data
* For females: pregnancy or lactation
* Women of childbearing potential (not postmenopausal or surgically sterile) not willing to use an effective method of contraception during the study. Effective methods are hormonal contraceptives (e.g., oral, implanted, or injected), intrauterine device (IUDs), and sexual abstinence.
* Patient committed to an institution by virtue of an order issued either by the courts or by an authority
* Patient who is unable to comply with the requirements of the study or who in the opinion of theinvestigator should not participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10-25 (Actual); Primary Completion 2016-04-14 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Freedom from aneurysm or dissection-related mortality | 30 days or less
  All deaths due to the treated pathology, including aneurysm rupture, complications of TEVAR leading to new aortic pathology (e.g., retrograde dissection leading to fatal cardiac tamponade).
Delivery and deployment success evaluation | 30 days or less
  Success will be based on the Delivery system evaluation, overall rate of vascular access complications
  * Rate of access failures
  * Rate of deployment system difficulties
  will be analyzed descriptively.

SECONDARY OUTCOMES:
Major device-related adverse events (MAE) | 30 days after the procedure
  MAEs include:
  * Endoleak (types I, Ill and IV)
  * Stent migration (>10 mm)2
  * Lumen occlusion
  * Aorta rupture
  * Conversion to open repair

CONTACTS AND LOCATIONS:
Overall Officials: Vicenç Riambau, Principal Investigator — Thorax Institute Hospital Clínic de Barcelona